CLINICAL TRIAL: NCT01303900
Title: Cardiovascular Disease in Adult Haemophilia Patients
Brief Title: Cardiovascular Disease (CVD) in Haemophilia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: UMC Utrecht (Other)
Responsible Party: Dr. E.P. Mauser-Bunschoten, Van Creveldkliniek, UMC Utrecht
Other Study IDs: CVD study 1
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Haemophilia; Cardiovascular Disease
Keywords: Haemophilia; Cardiovascular disease; Cardiovascular disease risk factors; Prospective; QRISK2; Hypertension; Hypercholesterolaemia; Diabetes; Obesity
MeSH Terms: conditions — Hemophilia A; Cardiovascular Diseases; Hypertension; Hypercholesterolemia; Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Life expectancy of hemophilia patients has improved considerably during the past decades and is approaching that of the general population. Hemophilia patients are therefore likely to be confronted with age-related disorders in addition to their primary illness and related diseases. Little is known about the occurrence of age-related co-morbidity, especially cardiovascular disease (CVD), in these patients. Low clotting factor levels are hypothesized to protect against both atherosclerosis and thrombus formation, resulting in a reduced risk of ischemic CVD. CVD mortality has been reported to be lower in haemophilia patients than in the general population, but data on non-fatal CVD are lacking, and no adjustment for CVD risk factors has been made so far.

The aim of our study is to assess the occurrence of CVD and its risk factors in a large cohort of haemophilia patients.

In this prospective multicenter cohort study in a group of 700-800 male patients with haemophilia A or B aged 30 years or older from The Netherlands and the UK, data on CVD history and CVD risk factors will be collected at baseline and compared with the general age-matched male population. Overall QRISK2 cardiovascular risk scores will be calculated and also compared with the general population. During a follow-up period of 5 and 10 years the occurrence of CVD events will be recorded and compared with the expected occurrence based on the QRISK2 scores and with data from the general population.

ELIGIBILITY:
Inclusion Criteria:

* Haemophilia A or B (mild, moderate or severe)
* Male gender
* Age 30 years or older
* Treated at participating haemophilia treatment center

Exclusion Criteria:

* No specific exclusion criteria

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All male haemophilia patients aged 30 years or older who are treated at one of the participating haemophilia treatment centers (Utrecht and Groningen, The Netherlands, and Sheffield, london, Cardiff and Glasgow, UK).
  Patients are recruited during regular clinic visits.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2009-01

PRIMARY OUTCOMES:
Ischemic cardiovascular disease | After 5 and 10 years
Cardiovascular disease risk factors | At baseline

SECONDARY OUTCOMES:
Association between clotting factor concentrate administration and cardiovascular events | 5-10 years

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (2):
  - Division of Haemostasis and Thrombosis, Department of Haematology, University Medical Center Groningen, Groningen
  - Van Creveldkliniek, University Medical Center Utrecht, Utrecht
- United Kingdom (4):
  - School of Medicine, Cardiff University and University Hospital of Wales, Cardiff
  - Glasgow Haemophilia and Thrombosis Centre, Royal Infirmary, Glasgow
  - Katharine Dormandy Haemophilia Centre and Haemostasis Unit, Royal Free Hospital, London
  - Sheffield Haemophilia and Thrombosis Centre, Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Derived] Van Der Valk P, Makris M, Fischer K, Tait RC, Chowdary P, Collins PW, Meijer K, van Vulpen LFD, Mauser-Bunschoten E, Schutgens REG. Reduced cardiovascular morbidity in patients with hemophilia: results of a 5-year multinational prospective study. Blood Adv. 2022 Feb 8;6(3):902-908. doi: 10.1182/bloodadvances.2021005260. PMID 34879394